CLINICAL TRIAL: NCT00747071
Title: Safety and Validation of Efficacy of Oral Administration of the Food Additive Colostrum Derived Anti Clostridium Difficile Antibodies
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsors decision
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Gadi Lalazar MD, Hadassah Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0180-08-HMO - CTIL
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2011-06

CONDITIONS: Clostridium Difficile-Associated Diarrhea
Keywords: Clostridium difficile; diarrhea; colostrum
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Hospitalized patients with Clostridium difficile associated diarrhea.
  Interventions: Drug: Colostrum
- 2 (Experimental): Close hospital contacts of each index case
  Interventions: Drug: Colostrum

INTERVENTIONS:
Drug: Colostrum — Daily administration of Colostrum derived antibodies against C. difficile.

SUMMARY:
This clinical study is designed to evaluate the safety and efficacy of oral administration of the food additive colostrum derived antibodies to Clostridium difficile for prevention of Clostridium difficile associated disease (CDAD).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Written informed consent
* At least 3 unformed or watery stools in each of the 2 previous 24 hour periods.
* Confirmed diagnosis of C. difficile associated diarrhea

Exclusion Criteria:

* Pregnant or breast feeding women
* Known allergy to milk or milk products
* Other etiology of diarrhea
* Active or Chronic conditions: IBD, short bowel syndrome, ischemic colitis Ileus
* Pseudomembranous colitis
* White blood count > 50,000
* Blood in stools
* Laxatives or motility drugs within 12 hours
* Inability to participate in adequate follow up
* Clinically unstable
* Investigator deems unsuitable
* Immune suppression (disease or treatment)
* GI surgery
* Past intestinal parasites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence of active Clostridium difficile associated diarrhea in index cases | 60 days
New cases of Clostridium difficile associated diarrhea in close hospital contacts. | 60 days

SECONDARY OUTCOMES:
Disease severity - duration, maximal intensity (number of stools) in index cases. | 60 days
Eradication of Clostridium difficile from stools | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel